CLINICAL TRIAL: NCT03627715
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Crossover Study Evaluating the Safety and Efficacy of Propagermanium in Patients With Diabetic Kidney Disease (DKD) Who Are Receiving Irbesartan
Brief Title: Safety and Effectiveness of Propagermanium in Diabetic Kidney Disease Participants Receiving Irbesartan
Acronym: ACTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dimerix Bioscience Pty Ltd (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMX-200-203 A; ACTRN12618000982213p (Registry Identifier: Australia New Zealand Clinical Trials Registry)
Record Dates: First submitted 2018-08-07; First posted 2018-08-13 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — propagermanium

STUDY DESIGN:
Intervention Model Description: Double-blind, Randomised, Placebo-Controlled, Crossover Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propagermanium then Placebo (Experimental): Propagermanium one capsule orally twice daily for 12 weeks. Compliance will be measured by drug accountability and completion of a participant diary.
  Participants will receive 12 weeks propagermanium and 12 weeks placebo separated by a 6 week washout period.
  Interventions: Drug: Propagermanium; Drug: Placebo
- Placebo then Propagermanium (Experimental): Propagermanium one capsule orally twice daily for 12 weeks. Compliance will be measured by drug accountability and completion of a participant diary.
  Participants will receive 12 weeks placebo and 12 weeks propagermanium separated by a 6 week washout period.
  Interventions: Drug: Propagermanium; Drug: Placebo

INTERVENTIONS:
Drug: Propagermanium — Immediate release capsule
  Other Names: PPG; repagermanium; DMX-200
Drug: Placebo — Placebo capsule

SUMMARY:
This study will be evaluating the safety and efficacy of propagermanium for the treatment of participants with DKD who are already taking irbesartan by:

* monitoring symptoms that participants may experience while on the study,
* measuring levels of protein in participant's urine and kidney function during the course of the study,
* measuring the levels of propagermanium and irbesartan that enters into participant's urine and blood, and
* comparing the propagermanium outcomes to participants' pre-study and placebo outcomes.

Eligible participants will randomly be assigned to one of two arms to receive both the propagermanium and placebo in different orders as follows, either:

Treatment Period 1 taking a propagermanium capsule twice a day for 12 weeks, followed by a six week washout period followed by Treatment Period 2 taking a placebo capsule twice a day for 12 weeks.

OR Treatment Period 1 taking a placebo capsule twice a day for 12 weeks, followed by a six week washout period followed by Treatment Period 2 taking a propagermanium capsule twice a day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 90 (inclusive) at screening;
2. A diagnosis of type 2 diabetes mellitus;
3. Baseline glycated haemoglobin (HbA1c) ≤ 12%;
4. Fasting plasma glucose < 21 mmol/L;
5. Must be receiving a stable dose of 300 mg daily of irbesartan (in any marketed formulation) for at least 3 months prior to screening, and have no plan to change treatment regime throughout the study;
6. Patients can be on stable doses of angiotensin converting enzyme inhibitors, aldosterone inhibitors, and/or sodium-glucose co-transporter-2 inhibitors. However, the dose and regimen must be stable for 3 months prior to screening and must have no plan to change treatment regime throughout the study;
7. Mean of two albumin creatinine ratio (ACR) values (screening and baseline) of more than or equal to 265 to 4,425 mg/g (30-500 mg/mmol) and within 30% of the screening value at the baseline assessment;
8. Estimated glomerular filtration rate more than or equal to 25-90 mL/min/1.73 m^2 using chronic kidney disease epidemiology collaboration (CKD-EPI) formula at screening;
9. Serum potassium levels (screening and baseline) less than 5.5 mmol/L. If either value is 5.5 or above the patient may receive dietary advice and be retested one week after the second value
10. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

    * Not of childbearing potential, defined as surgically sterile (documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or postmenopausal (no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone [FSH] level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.);
    * Of childbearing potential and agrees to use a highly effective method of contraception consistently during the treatment period and for at least 60 days after the last dose of investigational product;
11. A male patient with a female partner of childbearing potential is eligible to participate if he agrees to use acceptable contraception during the treatment period and for at least 60 days after the last dose of investigational product and refrains from donating sperm during this period;
12. Have given written informed consent prior to any study procedures being performed.

Exclusion Criteria:

1. A history of type 1 diabetes mellitus;
2. Current known non-diabetic renal disease. Patients with a history of other resolved renal diseases must be approved by the Sponsor;
3. A prior organ or stem cell transplant;
4. A major adverse cardiac event within 6 months before screening;
5. Patients receiving immunosuppressive medications including patients receiving > 5 mg prednisone;
6. Rapid estimated glomerular filtration rate decline with renal replacement likely during study
7. Lymphoma, leukaemia, or any malignancy within the past 5 years except for basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ that have been resected with no evidence of metastatic disease for 3 years;
8. Jaundice, active hepatitis, or known hepatobiliary disease (except asymptomatic cholelithiasis);
9. Alanine aminotransferase and/or aspartate aminotransferase more than two times the upper limit of normal at screening;
10. Participation in any clinical study with an experimental medication or device within 90 days or 5 half-lives (whichever is longer) of screening or have previously participated in a study involving propagermanium;
11. Positive screening assessment for viral hepatitis B surface antigen or hepatitis C virus (HCV) antibody AND positive HCV ribonucleic acid or human immunodeficiency virus (HIV);
12. Seated blood pressure of more than or equal to 160/100 mmHg at screening;
13. Body mass index more than or equal to 42 kg/m^2 at screening;
14. Past hospitalisation for a major depressive episode;
15. Is breast feeding or pregnant;
16. Unable to comply with the study procedures and assessments, including the ability swallow capsules;
17. Any other disease, physical or psychological condition that the investigator or sponsor believes may contraindicate the use of the investigational medicinal product or affect the interpretation of study results or render the patient at high risk from treatment complications;
18. Are investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
The Change in Albumin/Creatinine Ratio with Adjunct use of Propagermanium Compared to Placebo in Participants with DKD who are Receiving Irbesartan | Twelve weeks
  Assessed by measuring albumin/creatinine ratio.

SECONDARY OUTCOMES:
The Effect of Treatment with Propagermanium Compared to Placebo on Measures of Estimated Glomerular Filtration Rate | Twelve weeks
  Assessed by measuring estimated glomerular filtration rate.
The Number of Adverse Events with the Adjunct use of Propagermanium | Twelve weeks
  Adverse events will be recorded by a patient diary and by site staff during site visits.
The Effect of Treatment with Propagermanium on Measures of Proteinuria as measured by ACR | Eleven 24-hour urine samples at week -2, week -1, week 6, week 11, week 12.
  Assessed by measuring albumin/creatinine ratio at each end point.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Roger, MD, Principal Investigator — Renal Research
Locations (13):
- Australia (13):
  - Renal Research, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Boxhill Hospital, Box Hill, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Sunshine Hospital, Melbourne, Victoria
  - Melbourne Renal Research Group, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincents Hospital, Melbourne, Victoria
  - Epworth Hospital, Richmond, Victoria

IPD SHARING:
Plan to Share IPD: Undecided